CLINICAL TRIAL: NCT00352898
Title: Comparative Study Evaluating the Immunogenicity & Safety of MeMuRu-OKA Vaccine & Measles-mumps-rubella Vaccine (Priorix™) Co-administered With Varicella Vaccine (Varilrix™) in Children Primed With Both Measles-mumps-rubella & Varicella Vaccines
Brief Title: Immunogenicity, Safety of Measles-mumps-rubella-varicella Vaccine (MeMuRu-OKA) Compared to Priorix™ Given With Varilrix™
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 105909
Record Dates: First submitted 2006-07-14; First posted 2006-07-17 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Mumps; Rubella; Measles; Varicella
MeSH Terms: conditions — Mumps; Rubella; Measles; Chickenpox

INTERVENTIONS:
Biological: MeMuRu-OKA (study vac)
Biological: MMR, Varicella vacc (control)

SUMMARY:
Since measles-mumps-rubella (MMR) and varicella vaccinations are established as routine childhood practice and often co-administered during the second year of life, a combined measles-mumps-rubella-varicella (MeMuRu-OKA) vaccine is fully justified. Such a combined vaccine was developed and extensively studied in susceptible children. In countries where varicella mass-vaccination is already implemented, a transition period is necessary as children who started with separate first-dose vaccinations of MMR and varicella will receive a single shot of the combined vaccine as the second dose. To account for those situations, this study will evaluate the effect of the combined measles-mumps-rubella-varicella vaccine given in place of separate MMR and varicella vaccines as a second dose.

ELIGIBILITY:
Inclusion Criteria:

* Children must be healthy to participate

Exclusion Criteria:

* immunosuppressive (including HIV) conditions, allergic diseases, neurological disorders, known anaphylactic reaction to MMR vaccine, and fever (axillary temperature ³ 37.5°C at the time of vaccination) are excluding factors. Children must have received one dose (but not more) of MMR and of varicella vaccine at least 6 weeks before entering the study. They must not receive or have received other non-registered drug or vaccine within 30 days prior to study start, or immunosuppressants for more than 14 days. Immunoglobulins or any blood products are prohibited during the 6 months before and during the study, as well as vaccine other than that foreseen by the protocol, 30 days before until 56 days after vaccination. They must not have had measles, mumps, rubella or varicella, or have been exposed to those diseases within 30 days prior to study start. New-born infants (< 5 weeks of age), pregnant women without previous exposure to chickenpox, and immunodeficient persons cannot live in the same household as the vaccinated child.

Ages: 15 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2006-04; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Varicella, MMR titres at 42-56 days after first vaccination

SECONDARY OUTCOMES:
Seropositivity rates. Safety: solicited local/general, unsolicited AEs (42 days), SAEs (whole study)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Canada (3):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
- Italy (3):
  - GSK Investigational Site, Enna, Sicily
  - GSK Investigational Site, Ragusa, Sicily
  - GSK Investigational Site, San Gregorio Di Catania (CT), Sicily

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 105909 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 105909 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 105909 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 105909 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 105909 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 105909 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register